CLINICAL TRIAL: NCT03818815
Title: A Study to Assess the Safety, Tolerability and Efficacy of OP0201 as an Adjunct Treatment for Acute Otitis Media in Infants and Children Aged 6 to 24 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novus Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OP0201-C-006
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: OP0201 + Antibiotics (Active Comparator): OP0201 20mg per day+oral Amoxicillin-clavulanate in two divided doses for 10 days
  Interventions: Combination Product: OP0201; Drug: Amoxicillin-clavulanate
- Placebo Comparator: Placebo +Antibiotics (Placebo Comparator): Placebo 0 mg per day+oral Amoxicillin-clavulanate in two divided doses for 10 days
  Interventions: Combination Product: Placebo; Drug: Amoxicillin-clavulanate

INTERVENTIONS:
Combination Product: OP0201 — OP0201 20mg per day in two divided doses for 10 days
  Arms: Drug: OP0201 + Antibiotics
Combination Product: Placebo — Placebo 0mg per day in two divided doses for 10 days
  Arms: Placebo Comparator: Placebo +Antibiotics
Drug: Amoxicillin-clavulanate — Oral Amoxicillin-clavulanate in two divided doses for 10 days

SUMMARY:
The purpose of this study is to develop a better understanding of the safety, tolerability and efficacy of intranasal OP0201 as an adjunct treatment to oral antibiotics for the treatment of Acute Otitis Media (AOM) in infants and children.

ELIGIBILITY:
Inclusion Criteria includes but is not limited to:

1. Male and female infants and children aged ≥6 months to ≤24 months
2. Diagnosis of Acute Otitis Media (AOM) - moderate to severe bulging of the TM or mild bulging of TM and recent [less than 48 hours] onset of ear pain or intense erythema of the TM
3. Score of 5 or more on the 5 question version of AOM-SOS scale1
4. Written informed consent by the child's legal guardian and their willingness to ensure that study instructions are followed, all study-related visits are attended, that treatment administration is given, and Parent/Caregiver assessments are recorded according to the study protocol.
5. Intact tympanic membrane (TM) in both ears (e.g., no perforation)

Exclusion Criteria includes but is not limited to:

1. Allergy to penicillin or cephalosporin
2. History or presence of immunodeficiency disorders
3. Antimicrobial therapy within the 3 days (i.e., 72 hours) prior to Day 1
4. Craniofacial abnormalities (e.g., cleft palate or Down's Syndrome) that may interfere with Eustachian tube function
5. Disorders with decreased mucociliary clearance or higher viscosity of the mucous (e.g., cystic fibrosis, primary ciliary dyskinesia, Kartagener's syndrome)
6. Clinically relevant blockage of 1 or both nasal passages, as determined by the investigator's medical judgment

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital of Pittsburgh - General Academic Pediatrics Oakland Medical Building, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muniz GB, Shope TR, Bhatnagar S, Shaikh N, Haralam MA, Liu H, Martin JM, Pogoda JM, Hoberman A. Intranasal Surfactant for Acute Otitis Media: A Randomized Trial. Pediatrics. 2021 Dec 1;148(6):e2021051703. doi: 10.1542/peds.2021-051703. PMID 34851411
- See also: Related Info — http://novustherapeutics.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: OP0201 + Antibiotics: OP0201 20mg per day+oral Amoxicillin-clavulanate in two divided doses for 10 days
  OP0201 20mg per day+Amoxicillin-clavulanate: OP0201 20mg per day+oral Amoxicillin-clavulanate in two divided doses for 10 days
- Placebo Comparator: Placebo +Antibiotics: Placebo 0 mg per day+oral Amoxicillin-clavulanate in two divided doses for 10 days
  Placebo 0mg per day+Amoxicillin-clavulanate: Placebo 0mg per day+oral Amoxicillin-clavulanate in two divided doses for 10 days
Period: Overall Study
Arm/Group | Drug: OP0201 + Antibiotics | Placebo Comparator: Placebo +Antibiotics
Started | 56 | 47
Completed | 48 | 42
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo Comparator: Placebo + Antibiotics: Placebo 0 mg per day+oral Amoxicillin-clavulanate in two divided doses for 10 days
- Total: Total of all reporting groups
Arm/Group | Drug: OP0201 + Antibiotics | Placebo Comparator: Placebo + Antibiotics | Total
Number analyzed (Participants) | 56 | 47 | 103
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.4 (4.70) | 13.2 (5.01) | 13.3 (4.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 33 | 22 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 53 | 43 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 25 | 61
  White | 16 | 16 | 32
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: Days 1-28
Population: Subjects who received at least one intranasal spray of study treatment. Subjects will be summarized and analyzed based on treatment received. The number of participant analyzed differs from the number of participants assigned to each arm by 1 due to a protocol deviation of one subject assigned Active was inadvertently dosed with Placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: OP0201 + Antibiotics | Placebo Comparator: Placebo + Antibiotics
Number analyzed (Participants) | 55 | 48
Participants | 48 | 36

2. Primary Outcome: Evaluation of Efficacy (Otoscopy)
Description: Percentage of study participants with no bulging tympanic membrane
Time Frame: Day 4
Population: Subjects who were randomized excluding the first 3 subjects dosed (subject numbers 1001, 1002 and 1003), as there was a known device malfunction for these subjects. Subjects will be summarized and analyzed based on randomization assignment, regardless of treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Drug: OP0201 + Antibiotics | Placebo Comparator: Placebo + Antibiotics
Number analyzed (Participants) | 54 | 46
Percentage of participants | 51 | 47.3
Statistical Analysis 1: Comparison: Drug: OP0201 + Antibiotics vs Placebo Comparator: Placebo + Antibiotics; The summary statistics are based on subjects with non-missing data only; Test type: Superiority; p = 0.62, Regression, Logistic — The p-value was calculated using multiple imputation with number of imputations equal to percentage of missing data

3. Primary Outcome: Evaluation of Efficacy (Otoscopy)
Description: Percentage of study participants with no middle ear effusion
Time Frame: Day 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Drug: OP0201 + Antibiotics | Placebo Comparator: Placebo + Antibiotics
Number analyzed (Participants) | 54 | 46
Percentage of participants | 55.9 | 37.9
Statistical Analysis 1: Comparison: Drug: OP0201 + Antibiotics vs Placebo Comparator: Placebo + Antibiotics; The summary statistics are based on subjects with non-missing data only; Test type: Superiority; p = 0.07, Regression, Logistic — The p-value was calculated using multiple imputation with number of imputations equal to percentage of missing data

ADVERSE EVENTS:
Time Frame: 28 days
Description: The Safety Population analyzed includes all subjects who received at least one intranasal spray of study treatment. Subjects will be summarized and analyzed based on treatment received. The number of participant analyzed differs from the number of participants assigned to each arm by 1 due to a protocol deviation of one subject assigned Active was inadvertently dosed with Placebo.
Arm/Group | Drug: OP0201 + Antibiotics | Placebo Comparator: Placebo + Antibiotics
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/48
Other Adverse Events (participants affected / at risk) | 48/55 | 36/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: OP0201 + Antibiotics (N=55) | Placebo Comparator: Placebo + Antibiotics (N=48)
KAWASAKIS DISEASE (Vascular disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: OP0201 + Antibiotics (N=55) | Placebo Comparator: Placebo + Antibiotics (N=48)
Diarrhoea (Gastrointestinal disorders) | 24 (24) | 22 (23)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal Discharge Discolouration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 33 (39) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT03818815/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT03818815/SAP_001.pdf